CLINICAL TRIAL: NCT05291507
Title: A Feasibility Evaluation of the Muse Magnetic Resonance Guided Focused Ultrasound System
Brief Title: Feasibility Evaluation of the Muse Magnetic Resonance Guided Focused Ultrasound System
Acronym: BreastMRgFUS
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCI148669
Record Dates: First submitted 2022-03-02; First posted 2022-03-22 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: This is an open-label, single arm, single center, non-randomized feasibility study of the Muse MRgFUS System in subjects with breast cancer.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Muse MRgFUS System (Experimental): Subjects will undergo partial ablation of half (≤50%) of one of their tumors (if multifocal or multicentric disease) followed by surgical resection per standard of care.
  Interventions: Device: Muse MRgFUS System

INTERVENTIONS:
Device: Muse MRgFUS System — The intended use of the device is to thermally ablate breast tissue under magnetic resonance image guidance. The thermal ablation is performed non-invasively using extracorporeal focused ultrasound.

SUMMARY:
This is an open-label, single arm, single center, non-randomized feasibility study of the Muse MRgFUS System in subjects with breast cancer. Subjects will undergo partial ablation of half (≤50%) of one of their tumors (if multifocal or multicentric disease) followed by surgical resection per standard of care. The partial tumor ablation design will ensure that no information is lost that would impact the subject's standard of clinical care. Because current care often includes testing on the tumor, retaining a portion of viable tumor is advised by the clinical team. To ensure viable tissue confirmation, patients will be enrolled in two cohorts as described in the protocol. The investigators will use imaging correlation, histological evaluation, and subject reported outcomes to assess the safety, tolerability, and efficacy of the Muse MRgFUS System. This proposed study will adhere to the guidelines of subjects receiving a timely tumor resection after diagnosis. All subjects will undergo the definitive procedure of surgical resection per standard of care. Surgical resection cannot be delayed as a result of the ablation and should occur within 6 weeks after the decision to proceed with surgical resection. In cases where a surgery may occur outside of the 6 week window, prior approval from the external DSMC should be obtained. While MRgFUS ablation is designed to be a breast-conserving technique, the investigators will enroll patients that are undergoing any surgical resection, including both lumpectomy or mastectomy. Both surgical procedures will allow assessment of the defined primary, secondary and exploratory objectives.

ELIGIBILITY:
Inclusion Criteria:

* Subject is able to speak and understand English.
* Female subjects 18 years of age or older with invasive breast cancer undergoing surgery
* ECOG < 2.
* ASA (American Society of Anesthesiologists) Physical Status Classification Scale assessment of I-II.
* Adequate breast size for MUSE device assessed by physician prior to study enrollment.
* Able to provide informed consent and willing to sign an approved consent form that conforms to federal and institutional guidelines.
* Adequate Renal Function defined as an eGFR > 30 mL/min/1.73.
* Female subjects of childbearing potential must agree to use a highly effective method of contraception as described in Section 5.4.1.
* Negative pregnancy test or evidence of post-menopausal status or evidence of permanent surgical sterilization (i.e. bilateral oophorectomy, bilateral salpingectomy, or hysterectomy). The post-menopausal status will be defined as having been amenorrhoeic for 12 months without an alternative medical cause. The following age-specific requirements apply:

  * Women < 50 years of age:

    ---Amenorrhoeic for ≥ 12 months following cessation of exogenous hormonal treatments; and

    ----Luteinizing hormone and follicle-stimulating hormone levels in the post-menopausal range for the institution.
  * Women ≥ 50 years of age:

    * Amenorrhoeic for 12 months or more following cessation of all exogenous hormonal treatments; or
    * Had radiation-induced menopause with last menses >1 year ago; or
    * Had chemotherapy-induced menopause with last menses >1 year ago.

Exclusion Criteria:

* Receiving other investigational agents at the time of study registration.
* Prior systemic anti-cancer therapy or any investigational therapy for neoadjuvant treatment of breast cancer.
* Prior radiation therapy to the ipsilateral breast or radiation whose field(s) encompassed the breast within which the current diagnosis of cancer is made.
* The diagnosis of another malignancy within ≤ 2 years before study enrollment, except for those considered to be adequately treated with no evidence of disease or symptoms and/or will not require therapy during the study duration (i.e., basal cell or squamous cell skin cancer, carcinoma in situ of the breast, or bladder or of the cervix). Low risk malignancies may be allowed after discussion with PI and medical monitor.
* Women with breast implants
* Pregnant or lactating women
* Inability to lie prone for 90 minutes as reported by patient or determined by investigator assessment.
* Known prior adverse reaction or allergy to commonly used sedatives (i.e. versed, propofol) (NCI CTCAE v5.0 Grade ≥ 3).
* Known prior adverse reaction or allergy to gadolinium contrast (NCI CTCAE v5.0 Grade ≥ 3).
* Contraindication to MRI as determined by treating physician or patient response on MRI patient history and safety questionnaire (Appendix 4)
* Medical, psychiatric, cognitive, or other conditions in the opinion of the investigator that may compromise the subject's ability to understand the subject information, give informed consent, comply with the study protocol or complete the study.

Additional Exclusion Criteria for Cohort 1 patients only

* Patient's tumor is grade 3 as determined in consultation with pathologist and treating physician.
* The amount of invasive tumor in the core biopsy specimen is small as determined in consultation with pathologist and treating physician.
* Core biopsy result is equivocal for HER2 after testing by both in situ hybridization and immunohistochemistry.
* There is doubt about the handling of the core biopsy specimen (long ischemic time, short time in fixative, different fixative), or the test is suspected by the pathologist to be negative on the basis of testing error.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female subjects 18 years of age or older with unilateral, unifocal invasive breast cancer undergoing lumpectomy
Enrollment: 34 (Estimated)
Dates: Start 2023-01-23 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
frequency of adverse events (AEs), adverse device effects (ADEs), and serious adverse events (SAEs) characterized by type | 2 months
  evaluate the safety, feasibility, and tolerability of soft tissue ablation with the Muse MRgFUS system as assessed by subject-reported procedural pain and incidence of device- and procedure-related adverse device effects and adverse events
frequency of adverse events (AEs), adverse device effects (ADEs), and serious adverse events (SAEs) characterized by severity (as defined by the NCI CTCAE, version 5.0) | 2 months
  evaluate the safety, feasibility, and tolerability of soft tissue ablation with the Muse MRgFUS system as assessed by subject-reported procedural pain and incidence of device- and procedure-related adverse device effects and adverse events
frequency of adverse events (AEs), adverse device effects (ADEs), and serious adverse events (SAEs) characterized by seriousness | 2 months
  evaluate the safety, feasibility, and tolerability of soft tissue ablation with the Muse MRgFUS system as assessed by subject-reported procedural pain and incidence of device- and procedure-related adverse device effects and adverse events
frequency of adverse events (AEs), adverse device effects (ADEs), and serious adverse events (SAEs) characterized by duration | 2 months
  evaluate the safety, feasibility, and tolerability of soft tissue ablation with the Muse MRgFUS system as assessed by subject-reported procedural pain and incidence of device- and procedure-related adverse device effects and adverse events
frequency of adverse events (AEs), adverse device effects (ADEs), and serious adverse events (SAEs) characterized by relationship to the investigational intervention reported during and after the procedure as compared to baseline | 2 months
  evaluate the safety, feasibility, and tolerability of soft tissue ablation with the Muse MRgFUS system as assessed by subject-reported procedural pain and incidence of device- and procedure-related adverse device effects and adverse events

SECONDARY OUTCOMES:
Evaluate ablation efficacy by pathologic assessment | 1 month
  estimate ablation efficacy
Disease-free survival (DFS) as defined as the time from the date of ablation to the date of first recurrence or death from any cause | 5 years
  estimate disease-free survival (DFS) at 5 years post ablation
Overall survival (OS) as defined as the time from registration until death from any cause | 5 years
  estimate overall survival in this study population at 5 years post ablation
Evaluate ablation efficacy by MRI treatment assessment metrics of thermal dose | 1 month
  estimate ablation efficacy
Evaluate ablation efficacy by T1-weighted non-perfused volume. | 1 month
  estimate ablation efficacy

CONTACTS AND LOCATIONS:
Overall Officials: Cindy Matsen, MD, Principal Investigator — Huntsman Cancer Institute
Locations (1):
- Huntsman Cancer Institute at University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No